CLINICAL TRIAL: NCT03697668
Title: Triple Antimalarial Combination (Imatinib-DHA-PPQ) to Accelerate the Parasite Clearance and to Prevent the Selection of Resistant Parasites
Brief Title: Triple Antimalarial Combination to Accelerate the Parasite Clearance and to Prevent the Selection of Resistant Parasites
Acronym: Artesynib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nurex S.r.l. (Industry)
Collaborators: Università degli Studi di Sassari (Other); Purdue University (Other); Vinmec Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NUREX S.r.l
Record Dates: First submitted 2018-07-02; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Plasmodium Falciparum Malaria (Drug Resistant)
Keywords: Imatinib Mesylate; piperaquine phosphate; dihydroartemisinin
MeSH Terms: conditions — Malaria, Falciparum | interventions — Imatinib Mesylate; benzene-1,4-diphosphonic acid

STUDY DESIGN:
Intervention Model Description: interventional
Masking Description: The research method will be a Phase 2 trial, 2 arms, randomized, open label (only the microscopist will be blinded), adaptive, dose de-escalation, trial conducted in adult male subjects with uncomplicated P.falciparum malaria.
  In all phases, patients will be treated by a triple combination IMA-DHA-PPQ (ARM 1) or by the standard DHA-PPQ treatment (ARM 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- imatinib-Dihydroartemisinin-piperaquine (Experimental): triple combination
  Interventions: Drug: Imatinib
- Dihydroartemisinin-piperaquine (Active Comparator): standard of care
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Imatinib — triple combination for the treatment of malaria
  Other Names: Gleevec; Glivec
  Arms: imatinib-Dihydroartemisinin-piperaquine
Drug: Dihydroartemisinin-piperaquine — standard malaria treatment
  Other Names: Artekin; Eurartesim; Diphos; Timequin; Duocotecxin
  Arms: Dihydroartemisinin-piperaquine

SUMMARY:
The purpose of this study is to provide a new drug combination for a better treatment of P. falciparum for a faster parasite clearance and to counteract artemisinin resistance.

DETAILED DESCRIPTION:
According to WHO, resistance to artemisinin derivatives (ART) is emerging in many areas of the Greater Mekong Region as a delayed parasite clearance following a standard treatment by artemisinin combined therapy (ACT). Artemisinin resistance is often accompanied by the resistance to the partner drugs such as piperaquine (PPQ), mefloquine (MEF), amodiaquine (AQ) and lumefantrine (LF).

The slow and incomplete clearance of parasites following ACT treatment is considered to permit the selection of resistant parasites.

The availability of new, more efficient treatments accelerating the clearance of parasites is therefore needed to counteract the selection of ART resistant strains.

Imatinib (IMA) has been demonstrated to increase the efficacy of ART in a synergic fashion. This positive effect is further potentiated by low concentrations of PPQ.

IMA is active both on the intra-erythrocyte asexual forms and on gametocytes. It is therefore expected that the combination DHA-PPQ-IMA should lead to faster and radical clearance of the parasites, therefore reducing the frequency of healthy carriers and transmission.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with mild to moderate P. falciparum malaria
2. Adult male, age 18-55 years
3. Good health conditions other than malaria
4. The patient did not take anti-malarial drugs in the past 4 weeks

Exclusion Criteria:

1. unable to provide Informed Consent or Patient History Form
2. symptoms and signs of severe or complicated malaria including: continuous high fever over 39 °C, confusion, convulsions
3. parasitemia<150.000 parasites /microliter
4. other neurological or psychiatric symptoms or disorders
5. abnormal bleeding
6. resting hearth rate lower than 60 and higher than 100 bpm
7. abnormal ECG, history of cardiac diseases
8. male adults with corrected QT intervals > 450ms
9. signs, symptoms and laboratory results of impairment of vital organs such as liver, lungs, kidney and cardiovascular system
10. hemoglobin < 9.0 gm/100ml
11. symptoms and signs of infection such as pneumonia, dengue fever, and other viral or bacterial infection.
12. patients with symptoms of gastrointestinal infections or any sign of malabsorption that may interfere with drug absorption
13. concomitant infection by plasmodium species other than P. falciparum
14. inability to meet daily with local doctor during period of clinical trial
15. concomitant medicines like:

    1. medicines used to treat high cholesterol in the blood (such as atorvastatin, lovastatin, simvastatin);
    2. medicines used to treat hypertension and heart problems (such as diltiazem, nifedipine, nitrendipine, verapamil, felodipine, amlodipine);
    3. medicined used to treat HIV (antiretroviral medicines): protease inhibitors (such as amprenavir, atazanavir, indinavir, nelfinavir, ritonavir), non-nucleoside reverse transcriptase inhibitors (such as efavirenz, nevirapine);
    4. medicines used to treat microbial infections (such as telithromycin, rifampicin, dapsone);
    5. medicines used to help you fall asleep: benzodiazepines (such as midazolam, triazolam, diazepam, alprazolam), zaleplon, zolpidem;
    6. medicines used to prevent/treat epileptic seizures: barbiturates (such as phenobarbital), carbamazepine or phenytoin;
    7. medicines used after organ transplantation and in autoimmune diseases (such as cyclosporin, tacrolimus);
    8. sex hormones, including those contained in hormonal contraceptives (such as gestodene, progesterone, estradiol), testosterone; - glucocorticoids (hydrocortisone, dexamethasone); - omeprazole (used to treat diseases related to gastric acid production);
    9. paracetamol (used to treat pain and fever);
    10. theophylline (used to improve bronchial air flow);
    11. nefazodone (used to treat depression);
    12. aprepitant (used to treat nausea);

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-17 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Adverse Events | From baseline to day 42
  Occurrence of Adverse Events over 42 days observation period
Occurrence of Severe Adverse Events | From baseline to day 42
  Occurrence of Severe Adverse Events over 42 days observation period
Occurrence of Abnormal Physical Symptoms | From baseline to day 42
  Occurrence of Abnormal Physical Symptoms (Clinical Abnormalities) over 42 days observation period
Occurrence of Abnormal Laboratory Values | From baseline to day 42
  Occurrence of Abnormal Laboratory Values over 42 days observation period

SECONDARY OUTCOMES:
Frequency of residual parasitemia: % of patients with >1000 parasites/ ul at day 3 and 28 | day 3 and day 28
  Parasitemia is determined by assessing the parasite count in blood, using thin film, thick film and qPCR analysis.
Frequency of fever and malaria symptoms | day 3 and day 28
  Percentage of patients with fever or malaria symptoms observed at Phisical Visit at day 3 and 28.
Mean parasitemia in the control and investigational arms | day 2 and day 5
  Mean parasitemia by assessing the parasite count in blood, using thin film, thick film and qPCR analysis, expressed as parasites / ul at day 2, 3 and 5 measured in the control and investigational arms
Parasite half-life measured at 12 and 24 hours | from baseline to 24 hours post-treatment
  Mean parasite clearance half-life calculated using parasitemia measured at baseline, 12 and 24 hours post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Huynh D Chien, MD, PhD, Principal Investigator — UNIVERSITY OF HUE, VIETNAM AND VINMEC DANANG INTERNATIONAL HOSPITAL, Hai Chau, Danang.; Francesco M Turrini, MD, PhD, Principal Investigator — University of Turin, Italy
Locations (1):
- A Tuc, Hương Hóa, Quang Tri, Vietnam

IPD SHARING:
Plan to Share IPD: No